CLINICAL TRIAL: NCT02157948
Title: A Multicenter, Double-blind, Randomized Study to Assess the Efficacy and Safety of Denosumab Produced by Two Different Processes in Postmenopausal Women With Osteoporosis
Brief Title: A Double-blind Study to Assess the Efficacy and Safety of Denosumab Produced by Two Different Processes in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120187; 2013-001279-19 (EudraCT Number)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: Postmenopausal Osteoporosis
Keywords: postmenopausal osteoporosis; osteoporosis; postmenopausal; denosumab; women
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab CP2 (Active Comparator): Participants received 60 mg denosumab manufactured using the current CP2 process subcutaneously once every 6 months for 1 year.
  Interventions: Drug: Denosumab (CP2)
- Denosumab CP4 (Experimental): Participants received 60 mg denosumab manufactured using the new CP4 process subcutaneously once every 6 months for 1 year.
  Interventions: Drug: Denosumab (CP4)

INTERVENTIONS:
Drug: Denosumab (CP2) — Denosumab produced by a process referred to as CP2, administered subcutaneously from a prefilled syringe.
  Other Names: XGEVA®
  Arms: Denosumab CP2
Drug: Denosumab (CP4) — Denosumab produced by a process referred to as CP4, administered subcutaneously from a prefilled syringe.
  Arms: Denosumab CP4

SUMMARY:
This study will compare the effect of denosumab produced by two different manufacturing processes on bone mineral density at the lumbar spine in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to any study-specific activities/procedures
* Ambulatory postmenopausal women.
* Age 55 years or older
* Screening BMD value equivalent to a T-score less than or equal to -2.5 at the lumbar spine, total hip, or femoral neck.

Exclusion Criteria:

* Administration of osteoporosis treatments or bone active treatments within specific timeframes
* Vitamin D deficiency
* Diseases and conditions that affect bone metabolism (e.g., hypo/hyper-parathyroidism; hypo/hyperthyroidism, unless stable and well-controlled)
* Contraindications to denosumab therapy (e.g., hypocalcemia)

Ages: 55 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (10):
  - Research Site, Santa Maria, California
  - Research Site, South Lake Tahoe, California
  - Research Site, Lakewood, Colorado
  - Research Site, Gainesville, Georgia
  - Research Site, Bethesda, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Albuquerque, New Mexico
  - Research Site, Akron, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Duncansville, Pennsylvania
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Québec, Quebec
  - Research Site, Westmout, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Świdnik
  - Research Site, Warsaw

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 21 centers in Poland, Denmark, United States (US), and Canada. The first participant enrolled on 05 May 2014 and the last participant enrolled on 03 July 2014.
Pre-assignment Details: Ambulatory postmenopausal women 55 years or older with a bone mineral density (BMD) equivalent to a T-score of ≤ 2.5 at lumbar spine, total hip, or femoral neck were eligible to enroll.
  Five hundred and forty-seven women were screened; 394 were enrolled and 153 did not meet eligibility criteria.
Period: Overall Study
Arm/Group | Denosumab CP2 | Denosumab CP4
Started | 197 | 197
Received Treatment | 196 | 196
Completed | 188 | 188
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Specified Criteria | 2 | 1
Not completed — Decision by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab CP2 | Denosumab CP4 | Total
Number analyzed (Participants) | 197 | 197 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (6.8) | 68.3 (7.3) | 68.1 (7.0)
Age, Customized [Number; unit: participants]
  < 65 years | 65 | 70 | 135
  ≥ 65 years | 132 | 127 | 259
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 197 | 394
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 190 | 195 | 385
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Other | 1 | 0 | 1
Lumbar Spine Bone Mineral Density (BMD) Score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.75 (0.91) | -2.75 (0.75) | -2.75 (0.83)
Serum Type I Collagen C-telopeptide (CTX-1) [Median (Inter-Quartile Range); unit: ng/mL] | 0.433 [0.268 to 0.610] | 0.462 [0.328 to 0.641] | 0.452 [0.295 to 0.618]
Serum Procollagen Type 1 N-terminal Propeptide (P1NP) [Median (Inter-Quartile Range); unit: μg/L] | 56.6 [45.7 to 73.4] | 61.5 [45.1 to 75.6] | 59.3 [45.4 to 75.0]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine BMD
Description: Lumbar spine bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and Month 12
Population: The primary efficacy analysis subset included all randomized participants who had a baseline lumbar spine DXA BMD measurement and at least 1 postbaseline lumbar spine DXA BMD measurement. Postbaseline BMD values obtained at the early termination visit were carried forward as the month-12 value.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab CP2 | Denosumab CP4
Number analyzed (Participants) | 187 | 188
percent change | 5.78 (3.44) | 5.73 (3.08)
Statistical Analysis 1: Comparison: Denosumab CP2 vs Denosumab CP4; The treatment comparison was analyzed using the analysis of covariance (ANCOVA) model including treatment, baseline BMD value, machine type, and machine type-by-baseline BMD value interaction. The effect of denosumab CP4 on lumbar spine BMD at 12 months relative to the effect of denosumab CP2 was estimated by the least-squares mean of the treatment difference (denosumab CP4 - denosumab CP2) and the corresponding 2-sided 95% confidence interval (CI); Test type: Non-Inferiority or Equivalence — Non-inferiority Testing: The lower bound of the 2-sided 95% CI of the between-group difference (denosumab CP4 - denosumab CP2) in percent change from baseline in lumbar spine BMD at 12 months was compared with the non-inferiority margin of -1.44% for assessing non-inferiority; p < 0.001, ANCOVA — One-sided p-value based on the prespecified non-inferiority margin of -1.44% for lumbar spine; Difference from CP2 = -0.07, 95% CI 2-sided [-0.72 to 0.57]
Statistical Analysis 2: Comparison: Denosumab CP2 vs Denosumab CP4; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence Testing: The lower and upper bounds of the same 2-sided 95% CI of the between-group difference were compared with the equivalence margin of ±1.44% for assessing equivalence; p < 0.001, ANCOVA — Two-sided p-value based on the prespecified equivalence margin of ±1.44% for lumbar spine; Difference from CP2 = -0.07, 95% CI 2-sided [-0.72 to 0.57]

2. Secondary Outcome: Percent Change From Baseline in Serum Type I Collagen C-telopeptide (sCTX)
Time Frame: Baseline, month 1, month 6 and month 12
Population: The bone turnover marker (BTM) efficacy analysis subset includes all randomized participants who had a baseline measurement and at least one post baseline measurement. "n" indicates the number of participants with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Denosumab CP2 | Denosumab CP4
Number analyzed (Participants) | 196 | 193
percent change
  Month 1 (n = 195, 193) | -86.39 [-90.65 to -78.45] | -88.05 [-91.12 to -80.79]
  Month 6 (n = 191, 189) | -76.46 [-85.58 to -60.58] | -79.48 [-87.06 to -66.86]
  Month 12 (n = 187, 188) | -71.34 [-83.33 to -47.13] | -75.44 [-85.88 to -61.90]

3. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type 1 N-terminal Propeptide (P1NP)
Time Frame: Baseline, month 1, month 6 and month 12
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Denosumab CP2 | Denosumab CP4
Number analyzed (Participants) | 196 | 193
percent change
  Month 1 (n = 195, 193) | -29.59 [-38.06 to -20.02] | -29.86 [-38.80 to -20.90]
  Month 6 (n = 192, 190) | -76.63 [-82.90 to -66.69] | -77.74 [-85.02 to -70.31]
  Month 12 (n = 186, 188) | -71.44 [-77.64 to -57.35] | -72.08 [-80.24 to -62.40]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Denosumab CP2 | Denosumab CP4
Serious Adverse Events (participants affected / at risk) | 13/196 | 6/196
Other Adverse Events (participants affected / at risk) | 25/196 | 36/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab CP2 (N=196) | Denosumab CP4 (N=196)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab CP2 (N=196) | Denosumab CP4 (N=196)
Nasopharyngitis (Infections and infestations) | 15 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.